CLINICAL TRIAL: NCT00602758
Title: ART Adherence: Enhanced Counseling and Observed Therapy
Brief Title: Effectiveness of Enhanced Counseling and Observed Therapy on Antiretroviral Adherence in People With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH068197 (NIH); R01MH068197 (NIH); PA 01 0173; DAHBR 9A-ASGA
Record Dates: First submitted 2008-01-04; First posted 2008-01-28 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: AIDS; Adherence; Antiretroviral Therapy; HIV
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enhanced Counseling (Experimental): Participants meet with a counselor trained in motivational interviewing and cognitive behavioral techniques
  Interventions: Behavioral: Motivational interviewing with cognitive behavioral therapy
- Standard Care (No Intervention): Participants receive usual clinical care provided by health care providers and they participate only in evaluation components of the study
- Enhanced Counseling/Modified Directly Observed Therapy (Experimental): Participants receive their ART medications delivered to them by study staff and they receive the enhanced counseling
  Interventions: Behavioral: Motivational interviewing with cognitive behavioral therapy; Behavioral: Modified directly observed therapy

INTERVENTIONS:
Behavioral: Motivational interviewing with cognitive behavioral therapy — Counseling sessions are completed face-to-face or by telephone at baseline and Weeks 1, 2, 4, 6, 9, 11, 15, 19, and 23. Counselors are trained in motivational interview technique and focus on ART medication adherence.
  Other Names: Enhanced counseling (EC)
  Arms: Enhanced Counseling; Enhanced Counseling/Modified Directly Observed Therapy
Behavioral: Modified directly observed therapy — From baseline to Week 16, Monday through Friday, study staff meet the participants daily to observe one dose of their ART and to leave with the participants all other doses needed until the next observed dose. The frequency of observed doses begins to taper at Week 17 through to Week 24.
  Other Names: OT; Modified observed therapy (MDOT)
  Arms: Enhanced Counseling/Modified Directly Observed Therapy

SUMMARY:
This study will compare the effectiveness of enhanced counseling alone versus enhanced counseling combined with observed therapy at improving medication adherence in people with HIV.

DETAILED DESCRIPTION:
HIV is a virus that can lead to acquired immunodeficiency syndrome (AIDS), a disease that breaks down the immune system and allows for entry of life-threatening secondary infections. HIV is transmitted through the exchange of bodily fluids, primarily through sexual intercourse. Antiretroviral therapy (ART) has proven to be an effective treatment for inhibiting the replication of HIV, allowing for improved quality of life and survival. However, the long-term effectiveness of ART depends on strict adherence to a prescribed medication regimen. Previous studies have indicated that observing patients while they take their medications for a period of time can improve adherence to their prescribed drug regimens. This study will evaluate the effectiveness of enhanced counseling (EC) alone versus EC combined with modified directly observed therapy (mDOT) at improving medication adherence in people with HIV.

Participants in this 48-week study will be randomly placed into one of the following three treatment groups:

* Group 1 participants will receive standard care, which will involve the care that the clinic staff normally provide to all patients on HIV therapy.
* Group 2 participants will receive EC.
* Group 3 participants will receive EC with mDOT.

All participants will continue to take the anti-HIV medication regimen prescribed by their health care provider. However, participants will be asked to keep one medication type in a bottle that has a special Micro-Electro-Mechanical System (MEMS) cap. This electronic cap will record each time the participant opens the bottle. Participants will meet with study staff for MEMS cap data collection once weekly for the first 4 weeks, every 2 weeks up to Week 12, and then every 4 weeks thereafter.

EC will consist of 30- to 45-minute counseling sessions about medication adherence. Participants will meet in person with a counselor for the first five sessions, occurring at baseline and Weeks, 1, 2, 6, and 11. An additional five counseling sessions will be conducted by phone during Weeks 4, 9, 15, 19, and 23. Participants receiving mDOT will have their doses of HIV medication delivered to them by an mDOT worker for the first 24 weeks of treatment. Participants will select a time and location to meet with an mDOT staff member, who will then provide the daily doses of drugs and observe participants taking those drugs. Participants will meet with an mDOT worker 5 times a week from baseline to Week 16. Starting at Week 17, the number of weekly meetings will gradually taper until Week 24 when there will be no meeting and participants will return to obtaining and taking their HIV medications as done prior to study enrollment.

Evaluation visits will occur for all participants at baseline and Weeks 12, 24, 36, and 48. Evaluation sessions will last 45 minutes to 1 hour and will include questionnaires about adherence, knowledge and attitudes about HIV and HIV therapy, quality of life, support systems, health status, medical history, drug and alcohol use, and satisfaction with HIV care. Blood samples will also be taken to measure CD4 cell count and amount of virus in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Patient at participating clinical site
* English-speaking
* Initiating new ART (new or change in therapy) or nonadherent to ART as documented by care provider's assessment, patient self-report, and consistent HIV RNA laboratory results
* Lives within 45-mile radius of participating clinical site or able to participate in observed therapy procedures

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2004-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Adherence with ART as measured by Micro-Electro-Mechanical Systems (MEMS) | Measured at Week 48

SECONDARY OUTCOMES:
HIV RNA suppression | Measured at Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Goggin, PhD, Principal Investigator — University of Missouri, Kansas City
Locations (4):
- United States (4):
  - Kansas University Medical Center ID Clinic, Kansas City, Kansas
  - Truman Medical Center ID Clinic, Kansas City, Missouri
  - Kansas City Free Health Clinic, Kansas City, Missouri
  - Kansas City Veterans Administration Medical Center, Kansas City, Missouri

REFERENCES:
- [Background] Goggin K, Liston RJ, Mitty JA. Modified directly observed therapy for antiretroviral therapy: a primer from the field. Public Health Rep. 2007 Jul-Aug;122(4):472-81. doi: 10.1177/003335490712200408. PMID 17639650
- See also: Click here for more information on the Kansas City Adherence Study (MOTIV8) — http://cas.umkc.edu/psyc/motiv8/